CLINICAL TRIAL: NCT07079917
Title: Alveolar Ridge Augmentation Using Minimally Invasive Subperiosteal Tunneling With Xenogenic Bone Graft and Platelet-Rich Fibrin: Randomized Controlled Trial
Brief Title: Alveolar Ridge Augmentation Using Minimally Invasive Subperiosteal Tunneling With Xenogenic Bone Graft and PRF
Acronym: MISTT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Abanoub Maged Sobhy Morkos, Demonstrator at oral & maxillofacial department, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: will be ready at end of study
Record Dates: First submitted 2025-07-02; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- subperiosteal tunneling for horizontal alveolar ridge augmentation (Active Comparator): subperiosteal dissection through horizontal incision
  Interventions: Procedure: subperiosteal tunneling for horizontal alveolar ridge augmentation
- conventional surgical approach for horizontal alveolar ridge augmentation (Active Comparator): conventional full thickness trapezoidal flap for alveolar ridge augmentation
  Interventions: Procedure: conventional alveolar ridge augmentation

INTERVENTIONS:
Procedure: subperiosteal tunneling for horizontal alveolar ridge augmentation — subperiosteal dissection through horizontal incision only
  Arms: subperiosteal tunneling for horizontal alveolar ridge augmentation
Procedure: conventional alveolar ridge augmentation — horizontal alveolar ridge augmentation through trapezoidal flap
  Arms: conventional surgical approach for horizontal alveolar ridge augmentation

SUMMARY:
surgical horizontal augmentation for maxillary alveolar ridge using minimally invasive subperiosteal tunneling in comparison to conventional surgical technique

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old seeking an implant-supported restoration with deficient horizontal posterior maxillary alveolar ridge, at area of one or two missed teeth of less than 5 mm buccolingual width.
* Minimum vertical height of 8 mm.
* Gingival tissue of healthy adequate keratinization, more than 2mm.

Exclusion Criteria:

* The presence of uncontrolled diabetes or any other systemic condition which may complicate the surgical procedure or interfere with bone healing
* Radiotherapy to the head and neck region
* Chemotherapy within the last 12 months
* Uncontrolled periodontitis
* Smoking
* Bisphosphonate therapy
* Pregnancy
* Presence of periapical infection or lesion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-08-21 (Estimated); Study Completion 2026-06-21 (Estimated)

PRIMARY OUTCOMES:
Maxillary alveolar bone width | 6 months
  increase of the alveolar bone buccolingually for horizontal ridge augmentation

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt